CLINICAL TRIAL: NCT02690012
Title: Feasibility of Using an Integrated Consent Model to Compare Two Standard of Care Regimens for the Management of Hypomagnesemia From Anti-Cancer Therapies
Acronym: OTT 15-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20150853-01H
Record Dates: First submitted 2016-01-27; First posted 2016-02-24 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hypomagnesemia
MeSH Terms: interventions — Magnesium Oxide; magnesium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Magnesium oxide (Active Comparator): Participants will be given standard dose levels of Magnesium oxide according to the level of magnesium in blood.
  Interventions: Other: Magnesium Oxide
- Drug Magnesium citrate (Active Comparator): Participants will be given standard dose levels of Magnesium citrate according to the level of magnesium in blood.
  Interventions: Other: Magnesium Citrate

INTERVENTIONS:
Other: Magnesium Oxide — Magnesium Oxide
  Arms: Drug Magnesium oxide
Other: Magnesium Citrate — Magnesium Citrate
  Arms: Drug Magnesium citrate

SUMMARY:
Hypomagnesemia (hMg) is a common side effect of important anti-cancer therapies such as epidermal growth factor receptor inhibitors (EGFRIs) and platinum-containing anti-cancer drugs. EGFRIs, including cetuximab (cmab) and panitumumab (pmab), have been estimated to cause hMg in over 18% and 27% of patients respectively1, while 90% of patients receiving cisplatin will develop hMg if left untreated. The development of severe hMg may result in increased symptoms such as fatigue, neuromuscular changes, mental status changes and cardiac arrhythmias which could result in treatment delays and may compromise treatment efficacy. Despite the common occurrence of this toxicity, little is known regarding the optimal magnesium management strategy. As physicians do not know what the "best" treatment for patients is, genuine uncertainty ("clinical equipoise") exists. Physicians will choose between different "standards" of magnesium replacement in their personal practice, using idiosyncratic decision making processes, without the physician or the patient knowing the optimal option. This is not good for patients, physicians and society as a whole. Determining the optimal treatment remains an important medical issue for patients, physicians and society. This study will use a novel method to allow comparisons of established standard of care prophylactic treatment using the "integrated consent model" as part of a pragmatic clinical trial7. By integrating medical and clinical practices, physicians will be able to inform their patients about the randomized control trial, akin to a typical conversation between the physician and patient, without written informed consent. This clinical interaction would then be documented, as ordinarily done in practice. Medical and clinical practice will be intertwined with the patients' welfare at the forefront of our best interests.

ELIGIBILITY:
Inclusion Criteria:

* • Palliative-intent treatment with Cisplatin, Carboplatin, Panitumumab or Cetuximab and expected to receive ≥ 2 months of further therapy.

  * Potassium level within normal limits
  * Developed grade ≥1 hMg (Mg < lower limit of normal)
  * ECOG less than or equal to 2
  * ≥19 years of age
  * Able to swallow tablets/capsules
  * Able to provide verbal consent

Exclusion Criteria:

* baseline creatinine >1.5x upper limit of normal ULN
* Current use of oral or IV magnesium supplementation (patients who receive 1 gram of magnesium with their standard Cisplatin/Carboplatin chemotherapy regimens are eligible).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who are eligible and agree to participate in RCT. | one year
Percentage of medical oncologists who agree to participate in the study at study commencement and approach patients for the study. | one year

SECONDARY OUTCOMES:
Magnesium levels | One year
  Compare the differences in levels of magnesium between the two regimens
Cardiac risk | one year
  Determine whether systemic therapy-induced hypomagnesemia poses a serious risk of cardiac arrhythmias as measured by changes in average QTc intervals with changes in magnesium levels.
Cost factors | one year
  Determine cost differences between two magnesium replacement strategies.
Rates of treatment delays | one year
Rates of hospital admissions. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vickers, Dr., Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada